CLINICAL TRIAL: NCT00736424
Title: Brain Stimulation for Epilepsy Long Term Follow-up
Acronym: SUDEP
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: 1616
Record Dates: First submitted 2008-06-24; First posted 2008-08-15 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Epilepsy
Keywords: Epilepsy; SUDEP; DBS
MeSH Terms: conditions — Epilepsy; Sudden Unexpected Death in Epilepsy

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Have received bilateral AN stimulation of the anterior nucleus (AN) of the thalamus for epilepsy or are receiving it at the time of enrollment
  Interventions: Device: Itrel II™ and Soletra™ Epilepsy Control System

INTERVENTIONS:
Device: Itrel II™ and Soletra™ Epilepsy Control System — Bilateral neurostimulation of the anterior nucleus of the thalamus

SUMMARY:
The purpose of this study is to collect subject data to evaluate the rate of sudden unexplained death in epilepsy (SUDEP) with bilateral neurostimulation of the anterior nucleus of the thalamus in people diagnosed with refractory epilepsy. The data obtained from the physician initiated studies will be pooled with data collected in Medtronic-sponsored studies to assess SUDEP risk.

DETAILED DESCRIPTION:
Medtronic is conducting a pivotal clinical trial entitled Stimulation of the Anterior Nucleus of the Thalamus in Epilepsy (SANTÉ). One of the requirements of the SANTÉ study is to evaluate the rate of sudden unexplained death in epilepsy (SUDEP). Medtronic is aware of approximately 18 subjects with various types of epilepsy that have been treated with neurostimulation of the anterior nucleus of the thalamus outside the SANTÉ trial under five physician-sponsored studies. This protocol will initially collect information regarding the physician-sponsored study subjects' status. The goal of this study is to pool these data with the SANTÉ data for the purpose of estimating the SUDEP rate.

This is a multi-center, retrospective and prospective clinical study in patients previously implanted with devices that provide bilateral neurostimulation of the anterior nucleus of the thalamus during non-Medtronic-sponsored studies.

ELIGIBILITY:
Inclusion Criteria:

* Have received bilateral AN stimulation of the anterior nucleus of the thalamus (AN) for epilepsy or are receiving it at the time of enrollment
* For patients with therapy active at the time of enrollment, ability of the patient or legal representative to understand and provide signed consent for participating in the study
* For patients with therapy permanently discontinued or died at time of enrollment, the IRB/REB has approved a waiver allowing collection of the data OR the ability of the patient or legal representative to understand and provide signed consent/medical authorization

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will initially include five sites that conducted physician-sponsored studies in the US and Canada. Centers may be added as additional patients are identified.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The primary objective is to collect patient data that may be pooled with other data to estimate the SUDEP rate in people with refractory epilepsy receiving bilateral deep brain stimulation of the anterior nucleus of the thalamus. | 5 years (anticipated)

REFERENCES:
- See also: Related Info — http://www.epilepsycontrol.com